CLINICAL TRIAL: NCT04517617
Title: The Influence of Prenatal Factors Including Environment on Maternal Hemorrhage
Brief Title: The Influence of Prenatal Factors on Maternal Hemorrhage
Acronym: TIOPFOMH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: The First Affiliated Hospital of the Fourth Military Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2018LSK-245
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2021-08

CONDITIONS: Postpartum Hemorrhage
Keywords: pregnancy; prenatal factors; environment; genetics; hemoglobin; blood loss
MeSH Terms: conditions — Postpartum Hemorrhage; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples will be taken before and after childbirth to detect serum level of hemoglobin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The level of maternal air pollution exposure during pregnancy: The groups will be decided according to the level of maternal exposure to air pollution during pregnancy. Participants will be divided into experimental group (high level of maternal air pollution exposure) and control group (low level of maternal air pollution exposure) or other groups according to research and actual demand.
  Interventions: Other: The level of air pollution

INTERVENTIONS:
Other: The level of air pollution — The intervention measure is the level of air pollution, it is a non-human interventional measure based on the weighted average of various air pollutants monitored by air pollution monitoring stations during different period of pregnancy.he perinatal period.

SUMMARY:
This research evaluates the effects of prenatal factors on adverse pregnancy outcomes, the general demographic information, the level of maternal exposure to air pollution, the environmental condition, pregnancy-related information, the occurrence of adverse pregnancy outcomes, and serum indicators of pregnant women during pregnancy are collected. Finally, the research explores that whether prenatal factors including environment can mediate the occurrence of maternal hemorrhage.

DETAILED DESCRIPTION:
The degree of hemoglobin changes before and after delivery can be used as an index, to accurately estimate postpartum hemorrhage in clinical practice. Postpartum hemorrhage is the leading cause of maternal death in the world, accounting for 30% of maternal deaths. Studies have shown that most deaths caused by postpartum hemorrhage are avoidable. Domestic and foreign literature reports that the incidence of postpartum hemorrhage is 5%~10%, however, the amount of blood loss clinically estimated is often lower than the actual amount, the actual incidence of postpartum hemorrhage is higher. A large number of studies have confirmed that maternal exposure to air pollution during pregnancy such as particulate matter (PM), nitrogen dioxide (NO2), sulfur dioxide (SO2), ozone (O3), carbon monoxide (CO) can increase the risk of adverse pregnancy outcomes, including miscarriage, gestational diabetes mellitus(GDM), hypertensive disorder complicating pregnancy, preterm birth and low birth weight(LBW). So, a prospective cohort study is conducted to explore the influence of prenatal factors and environment on maternal hemorrhage.

Research content: This research is a prospective cohort study from June 2020 to December 2022, 500 pregnant women will be recruited from the First Affiliated Hospital of Xi'an Jiaotong University and First Affiliated Hospital of the Fourth Military Medical University. A health management birth cohort will be established. ①To construct a spatial and temporal series about maternal hemorrhage influenced by maternal exposure to air pollution during pregnancy; ②To explore the effects of prenatal factors and environment on maternal hemorrhage.

Research meaning：① Practical significance: To explore the factors that affect maternal hemorrhage, and to reduce the occurrence of postpartum hemorrhage, which contributes to reducing the healthy risks and medical economic burdens caused by the healthy problems of mothers and children. ② To define the critical period of the developing of maternal hemorrhage in spatial and temporal series, and to calculate the cutoff value of air pollution on maternal hemorrhage, propose short-term control target of air pollution related to maternal and child health, construct the first-level prevention strategy for adverse pregnancy outcomes.

Research steps: ① Complete the recruiting of subjects, which meet the inclusion and exclusion criteria sign an informed consent before the carrying out of research; ② Follow up: Questionnaires will be conducted to acquire the information including sociodemographic characteristics, menstrual history and childbearing history, residence during pregnancy, lifestyle and diet habits, the information of illness and medication, history of past illness, etc. Then the maternal exposure level of air pollutants in every trimester will be calculated, based on air pollution detection station, from Shaanxi Meteorological and Environment Bureau according to residence information of participants; ③ Serum indicators: fasting venous blood samples will be taken before and after childbirth to detect serum level of hemoglobin, all the blood samples will be taken and tested in the laboratory of the First Affiliated Hospital of Xi'an Jiaotong University and First Affiliated Hospital of the Fourth Military Medical University; ④ Monitoring of postpartum hemorrhage: closely monitor the volume of blood loss. During the whole study period, the subjects could withdraw the cohort at any time.

Prenatal hemoglobin level: blood hemoglobin level within one week before delivery; Postpartum hemoglobin level: blood hemoglobin level 1 day after delivery; The difference of hemoglobin before and after delivery: prenatal hemoglobin level minus postpartum hemoglobin level (if he patient received red blood cell transfusion during this period, this value is the degree of hemoglobin change after calibration); The 24 h postpartum hemorrhage is calculated as 400 ml for every 10g/L drop in hemoglobin; Birth weight: the weight of newborn within the first hour.

Statistical method: ①Univariate analysis: The maternal exposure levels of air pollution during pregnancy will be treated as independent variables, postpartum hemorrhage will be treated as dependent variables, univariate logistic regression will be used to analyze the relationship between them; ②Multivariate analysis: postpartum hemorrhage will be taken as dependent variables, maternal exposure levels, sociodemographic characteristics, nutritional status, dietary status, and other factors are included as independent variables, the multivariate logistic regression analysis will be used to data analysis. In the multivariate regression the odds ration value and 95% confidence intervention of air pollution to affect adverse pregnancy outcomes will be calculated adjusted for sociodemographic characteristics, nutrition, dietary conditions and other factors; ③Spatial and temporal series analysis will be adapted to define the critical period of the developing of postpartum hemorrhage under maternal exposure to air pollution, and calculate the cut-off value of air pollution about postpartum hemorrhage.

Research planning: ①Complete research design, follow-up questionnaires, and pre-experiments before July 2020; ②Complete enrollment of subjects, collect pregnancy-related information, follow-up of the study subjects, detecting of serum indicators, monitor the occurrence of postpartum hemorrhage before July 2022; ③Complete data export and analysis about basic information and data analysis; ④Clarify the relationship between maternal air pollution exposure during pregnancy and postpartum hemorrhage, explore the potential mechanism in the occurrence of postpartum hemorrhage influenced by prenatal factors and environment.

ELIGIBILITY:
Inclusion Criteria:

* The Pregnant women gave birth in the First Affiliated Hospital of Xi'an Jiaotong University and First Affiliated Hospital of the Fourth Military Medical University;
* This pregnancy is natural conception, the last menstrual period is definite and the menstrual cycle is basically regular;
* The pregnant women volunteer to participate in this study and sign the informed consent.

Exclusion Criteria:

* The pregnant women have placental abruption;
* The pregnant women have placenta previa;
* The pregnant women have placental implantation;
* The pregnant women have placental abruption;
* The pregnant women with incomplete clinical records.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study participants are healthy pregnant women from the First Affiliated Hospital of Xi'an Jiaotong University and First Affiliated Hospital of the Fourth Military Medical University, who meet the inclusion and exclusion criteria, and sign the informed consent before the implementation of this research.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The Influence of Prenatal Factors Including Environment on Maternal Hemorrhage. | Prenatal hemoglobin level: blood hemoglobin level within one week before delivery; Postpartum hemoglobin level: blood hemoglobin level 1 day after delivery
  The 24 h postpartum hemorrhage is calculated as 400 ml for every 10g/L drop in hemoglobin; The difference of hemoglobin before and after delivery: prenatal hemoglobin level minus postpartum hemoglobin level (if he patient received red blood cell transfusion during this period, this value is the degree of hemoglobin change after calibration);

CONTACTS AND LOCATIONS:
Overall Officials: Wenfang Yang, Ph.D, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No